CLINICAL TRIAL: NCT06119061
Title: Telavancin Blood and Cerebrospinal Fluid Concentrations in Patients With External Ventricular Drainage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aaron Cook (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Aaron Cook, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 84795
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: pharmacokinetics; augmented renal clearance
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telavancin (Experimental): Subjects receiving telavancin for pharmacokinetic sampling
  Interventions: Drug: Telavancin Injection

INTERVENTIONS:
Drug: Telavancin Injection — Telavancin 10mg/kg (maximum 1000mg) administered intravenously over 60 minutes (through a central venous catheter whenever available).
  Other Names: Vibativ

SUMMARY:
The proposed study aims to evaluate the CNS penetration of telavancin in a critically ill population using cerebrospinal fluid (CSF) drawn from external ventricular drains (EVDs). Patients with EVDs were chosen as the target population because they frequently require prolonged admission to the intensive care unit and drainage of CSF in order to prevent hydrocephalus. The estimated sample size is 20 subjects. This is a prospective cohort of patients with SAH. Patients will be included if they have an in-dwelling EVD, aged 18-85 years old.

Subjects will receive telavancin 10mg/kg (maximum 1000mg) every 24 hours for 3 consecutive doses. Serial serum and CSF samples will be obtained. An 8-hour urine collection will be completed on study day 2 in order to define the patient's measured creatinine clearance.

DETAILED DESCRIPTION:
Telavancin exhibits potent and durable activity against target pathogens for bacterial meningitis and ventriculitis. There is a potential role for telavancin in treating Gram positive CNS pathogens, particularly in patients with resistant pathogens or in those who are intolerant to other commonly used antimicrobials. The proposed study aims to evaluate the CNS penetration of telavancin in a critically ill population using cerebrospinal fluid (CSF) drawn from external ventricular drains (EVDs) in patients who have had spontaneous subarachnoid hemorrhage (SAH). Patients with SAH were chosen as the target population because they frequently require prolonged admission to the intensive care unit and drainage of CSF in order to prevent hydrocephalus. The estimated sample size is 15 subjects.

Methods: This is a prospective cohort of patients with SAH. Patients will be included if they have a spontaneous SAH, aged 18-65 years old, Hunt-Hess score of 1-4 & has an actively draining ventriculostomy. Patients will be excluded if they have a history of telavancin or similar agents, reduced renal function (estimated creatinine clearance < 50ml/min) at the time of consent, severe anemia (hemoglobin < 7gm/dl), vulnerable population (pregnant, prisoner).

Subjects will receive telavancin 10mg/kg (maximum 1000mg) every 24 hours for 3 consecutive doses. Baseline serum and CSF samples will be drawn before the initial dose of telavancin. Serial serum and CSF samples will be obtained after the first and third doses (1, 3, 6, 23 hours after infusion). A terminal concentration will also be obtained approximately 48 hours after the last dose. An 8-hour urine collection will be completed on study day 2 in order to define the patient's measured creatinine clearance.

Major Goals Goal 1. Determine the CNS penetration of telavancin in critically ill patients with SAH. Serial CSF and serum samples will be obtained from SAH patients with EVDs before and after scheduled telavancin doses in order to determine the degree of CNS penetration of telavancin.

Goal 2. Describe the pharmacokinetics of telavancin in critically ill patients with SAH. Patients with SAH frequently exhibit augmented renal clearance.(5) This increase in renal clearance has been demonstrated to affect the pharmacokinetics of numerous renally-eliminated medications. Volume of distribution may also be affected for many medications (such as telavancin) due to the frequent aggressive measures needed to maintain euvolemia or hypervolemia in some instances (due to SAH-induced vasospasm) and changes in serum albumin concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-85 years
* Actively draining ventriculostomy

Exclusion Criteria:

* history of hypersensitivity to telavancin or similar agents
* reduced renal function (estimated creatinine clearance < 50/ml) at the time of consent
* severe anemia (hemoglobin < 7gm/dl)
* vulnerable population (pregnant, prisoner)
* concomitant antimicrobial therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the CNS penetration of telavancin in critically ill patients with External Ventricular Drainage | 3 days
  Telavancin concentrations in CSF drawn from external ventricular drains will be compared to samples from the serum to determine the degree to which telavancin is present in the CNS

SECONDARY OUTCOMES:
Describe the pharmacokinetics of telavancin in critically ill patients with External Ventricular Drainage | 5 days
  Analyze serial serum concentrations of telavancin to determine the population's clearance, half-life, & volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Aaron M Cook, PharmD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Data from this study may be requested from other researchers 2 years after the completion of the primary endpoint by contacting the primary investigator

REFERENCES:
- [Background] Tunkel AR, Hasbun R, Bhimraj A, Byers K, Kaplan SL, Scheld WM, van de Beek D, Bleck TP, Garton HJL, Zunt JR. 2017 Infectious Diseases Society of America's Clinical Practice Guidelines for Healthcare-Associated Ventriculitis and Meningitis. Clin Infect Dis. 2017 Mar 15;64(6):e34-e65. doi: 10.1093/cid/ciw861. PMID 28203777
- [Background] Thigpen MC, Whitney CG, Messonnier NE, Zell ER, Lynfield R, Hadler JL, Harrison LH, Farley MM, Reingold A, Bennett NM, Craig AS, Schaffner W, Thomas A, Lewis MM, Scallan E, Schuchat A; Emerging Infections Programs Network. Bacterial meningitis in the United States, 1998-2007. N Engl J Med. 2011 May 26;364(21):2016-25. doi: 10.1056/NEJMoa1005384. PMID 21612470
- [Background] Rybak MJ, Le J, Lodise TP, Levine DP, Bradley JS, Liu C, Mueller BA, Pai MP, Wong-Beringer A, Rotschafer JC, Rodvold KA, Maples HD, Lomaestro B. Therapeutic Monitoring of Vancomycin for Serious Methicillin-resistant Staphylococcus aureus Infections: A Revised Consensus Guideline and Review by the American Society of Health-system Pharmacists, the Infectious Diseases Society of America, the Pediatric Infectious Diseases Society, and the Society of Infectious Diseases Pharmacists. Clin Infect Dis. 2020 Sep 12;71(6):1361-1364. doi: 10.1093/cid/ciaa303. PMID 32658968
- [Background] Cook AM, Hatton-Kolpek J. Augmented Renal Clearance. Pharmacotherapy. 2019 Mar;39(3):346-354. doi: 10.1002/phar.2231. Epub 2019 Mar 11. PMID 30723936
- [Background] Carrie C, Bentejac M, Cottenceau V, Masson F, Petit L, Cochard JF, Sztark F. Association between augmented renal clearance and clinical failure of antibiotic treatment in brain-injured patients with ventilator-acquired pneumonia: A preliminary study. Anaesth Crit Care Pain Med. 2018 Feb;37(1):35-41. doi: 10.1016/j.accpm.2017.06.006. Epub 2017 Jul 26. PMID 28756331
- [Background] Shaw JP, Seroogy J, Kaniga K, Higgins DL, Kitt M, Barriere S. Pharmacokinetics, serum inhibitory and bactericidal activity, and safety of telavancin in healthy subjects. Antimicrob Agents Chemother. 2005 Jan;49(1):195-201. doi: 10.1128/AAC.49.1.195-201.2005. PMID 15616296
- [Result] Albanese J, Leone M, Bruguerolle B, Ayem ML, Lacarelle B, Martin C. Cerebrospinal fluid penetration and pharmacokinetics of vancomycin administered by continuous infusion to mechanically ventilated patients in an intensive care unit. Antimicrob Agents Chemother. 2000 May;44(5):1356-8. doi: 10.1128/AAC.44.5.1356-1358.2000. PMID 10770777
- [Result] Stucki A, Gerber P, Acosta F, Cottagnoud M, Cottagnoud P. Efficacy of telavancin against penicillin-resistant pneumococci and Staphylococcus aureus in a rabbit meningitis model and determination of kinetic parameters. Antimicrob Agents Chemother. 2006 Feb;50(2):770-3. doi: 10.1128/AAC.50.2.770-773.2006. PMID 16436742